CLINICAL TRIAL: NCT06105892
Title: Eye Recovery Automation for Post Injury Dysfunction
Brief Title: Eye Recovery Automation for Post Injury Dysfunction (iRAPID)
Acronym: iRAPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Jersey Institute of Technology (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); University of New Mexico (Other); Biomedical Research Institute of New Mexico (Other); New Mexico VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chang Yaramothu, Assistant Professor, New Jersey Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SQRL001; W81XWH22C0146 (Other Grant/Funding Number: U.S. Army Medical Research and Development Command)
Record Dates: First submitted 2023-10-17; First posted 2023-10-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Convergence Insufficiency; Traumatic Brain Injury; Concussion, Mild
Keywords: Virtual Reality; Cross-Sectional; Therapy; Convergence Insufficiency; Traumatic Brain Injury
MeSH Terms: conditions — Ocular Motility Disorders; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Each of these participant cohorts (Control and TBI with CI [PTCI]) will be randomly halved to generate a total of four cohorts for a semi-crossover study design: 1) BNC Active, 2) BNC Sham [Placebo], 3) PTCI Active, and 4) PTCI Sham [control group]. PTCI participants in Sham will later undergo active therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the clinical coordinators and technicians (programming the therapy) will know the therapy type. Investigators, clinical examiners, and data analysts, will be masked to therapy type until performing group level analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- BNC Active (Experimental): Binocularly normal controls receiving active therapy
  Interventions: Device: Virtual Eye Rotation Vision Exercise (VERVE)
- BNC Sham (Sham Comparator): Binocularly normal controls receiving sham therapy
  Interventions: Device: Sham VR Therapy
- PTCI Active (Experimental): Post-traumatic Convergence Insufficiency participants receiving active therapy
  Interventions: Device: Virtual Eye Rotation Vision Exercise (VERVE)
- PTCI Sham (Sham Comparator): Post-traumatic Convergence Insufficiency participants receiving sham therapy
  Interventions: Device: Sham VR Therapy

INTERVENTIONS:
Device: Virtual Eye Rotation Vision Exercise (VERVE) — VERVE utilizes a virtual reality (VR) headset with integrated eye-tracking where the patient makes specific vergence eye movements by playing a VR game controlled by eye movements. Participants will be making convergence and divergence eye movements as steps and ramps.
  Other Names: Virtual Reality Vergence Exercises; Vergency Therapy
  Arms: BNC Active; PTCI Active
Device: Sham VR Therapy — VERVE game without changes in eye movement demands. Maximizing gameplay with no intervention.
  Arms: BNC Sham; PTCI Sham

SUMMARY:
This study will test a portable virtual reality (VR) system with integrated eye tracking called Virtual Eye Rotation Vision Exercises (VERVE). The proposed VERVE platform will deliver vergence therapy in an automated manner. This research will involve 30 non-traumatic brain injury (TBI) binocularly normal (BNC) Veterans and 50 post-traumatic convergence insufficiency (PTCI) Veterans who will undergo Active and Sham therapy (equally divided groups) to determine the effectiveness of VERVE vergence therapy.

ELIGIBILITY:
Mild Traumatic Brain Injury (mTBI) Cohort Inclusion Criteria:

1. are aged 18 - 40;
2. have suffered a mTBI according to VA/Department of Defense (DoD) criteria with documented evidence of alteration of consciousness (AOC) < 24 hours or loss of consciousness (LOC) less than 30 minutes;
3. were injured between 1 month and 15 years ago;
4. received a Glasgow coma scale (GCS) score of between 13 and 15 upon emergency department (ED) admission, if available;
5. experienced less than 24 hours of post-traumatic amnesia (PTA), if any;
6. have ongoing post-concussive symptoms as evidenced by a score of 18 or greater or a score of 2 or greater on question 6 (vision problems, blurring, trouble seeing) on the Neurobehavioral Symptom Inventory (NSI);
7. have ongoing vision-related symptoms as evidenced by a score of 31 or higher on the Brain Injury Vision Symptom Survey (BIVSS);
8. have PTCI as evidenced by obtaining a score of 21 or higher on the convergence insufficiency symptom survey (CISS), a specific measure of convergence insufficiency;
9. are fluent in English; and
10. have been on stable doses of any vision-altering medications for the past 2 months.
11. Stereopsis of 500 sec arc using Randot Stereo Test.
12. Exophoria at near 4 prism-diopter (PD) or greater than magnitude at distance
13. Near point of convergence (NPC) > 5 cm
14. Convergence amplitude at near < 15PD break or the Sheard criterion not met

Control Inclusion Criteria:

1. are aged 18 - 40;
2. CISS score of 20 or lower;
3. near point of convergence (NPC) < 6cm; and
4. positive fusional range >15 prism diopters.
5. Stereopsis of 500 sec arc using Randot Stereo Test.

Exclusion Criteria:

1. prior history of other neurological diseases, so as to reduce the risk of confounding effects on vision;
2. history of psychosis, as there are known visual performance findings associated with psychosis;
3. history of current or recent (within two years) substance/alcohol dependence, to reduce confounding effects on visual function
4. recent medical hospitalization (within three weeks), to reduce risk of rehospitalization during the study;
5. any condition that would prevent the participant from completing the protocol;
6. appointment of a legal representative, to avoid coercion of a vulnerable population;
7. any ongoing litigation related to TBI, to prevent interference with legal proceedings;
8. membership in an identified vulnerable population, including minors and prisoners, so as to prevent coercion.
9. Previous vergence therapy, orthoptics, home-based therapy, etc.
10. Amblyopia or constant strabismus or strabismus surgery.
11. High refractive error: Myopia ≥ 6.0PD sphere; Hyperopia ≥ 5.0PD sphere; Astigmatism ≥ 4.0PD; Anisometropia >1.5PD difference between eyes; Prior refractive surgery.
12. Manifest or latent nystagmus evident clinically.
13. Systemic diseases that affect accommodation, vergence, or ocular motility (i.e. multiple sclerosis, Graves' thyroid disease, myasthenia gravis, diabetes, chemotherapy or Parkinson disease).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Near Point of Convergence | Baseline (preintervention), within 1 week after session 4 of intervention, within 1 week after session 8 of intervention, within 1 week after session 12 of intervention, and within 1 week after intervention
  Normal range is < 6 cm
Positive Fusional Vergence | Baseline (preintervention), within 1 week after session 4 of intervention, within 1 week after session 8 of intervention, within 1 week after session 12 of intervention, and within 1 week after intervention
  Normal range is >15 Prism Diopters
Objective Eye-Tracking Measures (Peak Velocity) | Baseline (preintervention) and within 1 week after intervention
  measured in degress/second
Objective Eye-Tracking Measures (Response Accuracy) | Baseline (preintervention) and within 1 week after intervention
  measured as a percentage of response divided by target amplitude

SECONDARY OUTCOMES:
Brain Injury Vision Symptom Survey | Baseline (preintervention) and within 1 week after intervention
  Normal range is < 31 for adults
Neurobehavioral Symptom Inventory | Baseline (preintervention) and within 1 week after intervention
  Normal range is < 18 for adults
Convergence Insufficiency Symptom Survey | Baseline (preintervention) and within 1 week after intervention
  Normal range is < 21 for adults

CONTACTS AND LOCATIONS:
Overall Officials: Chang Yaramothu, PhD, Principal Investigator — New Jersey Institute of Technology
Locations (1):
- New Mexico VA Health Care System, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on Federal Interagency Traumatic Brain Injury Research Informatics System (FITBIR).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: On an annual basis after the start of the study and at the conclusion of the study